CLINICAL TRIAL: NCT01871935
Title: Comparison of the Effects of Atropine on Haemodynamics and Tissue Oxygenation in Anaesthesia With Propofol and Sufentanil Versus Propofol and Remifentanil
Brief Title: Atropine Effects in Anaesthesia With Sufentanil vs. Remifentanil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, A.F.Kalmar, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SuRe-002
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Haemodynamic Fluctuations During Off-pump CABG.
MeSH Terms: interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Active Comparator): Anaesthesia with remifentanil/propofol
  Interventions: Drug: Remifentanil
- Sufentanil (Active Comparator): Anaesthesia with sufentanil/propofol
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Remifentanil — Anaesthesia with remifentanil/propofol.
  Arms: Remifentanil
Drug: Sufentanil — Anaesthesia with sufentanil/propofol
  Arms: Sufentanil

SUMMARY:
Induction of general anaesthesia with a combination of opiates and hypnotics often induces vasodilation resulting in several haemodynamic effects such as a decrease in blood pressure (MAP), heart rate (HR) and cardiac output (CO). This haemodynamic suppression may jeopardize tissue oxygenation, particularly cerebral oxygenation. Previous research of the investigators group has revealed that atropine has an exceptionally beneficial effect on the determinants of tissue oxygen delivery as well as on tissue oxygenation. The investigators have demonstrated a significant and clinically relevant increase in CO and cerebral tissue oxygenation (SctO2) for a desired increase in MAP. This is in steep contrast with the more usual clinical practice of administrating classical vasoactive medication such as phenylephrine or norepinephrine, since the two latter have an even negative effect on CO and SctO2. In previous research the investigators used standardized target controlled propofol/remifentanil infusions for induction and maintenance of anaesthesia. It is known that remifentanil has more intense haemodynamic side-effects compared to other opiates such as fentanyl, sufentanil or alfentanil. This raises the question whether the beneficial effect of atropine is restricted to propofol/remifentanil anaesthesia, or if this is equally valid during anaesthesia of propofol combined with other opiates such as sufentanil.

Patients undergoing off-pump coronary artery bypass grafting (CABG) require a long and deep general anaesthesia, which is usually performed with the combination of drugs as mentioned above. Because these patients often experience severe haemodynamic fluctuations they need to be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older.
* Elective CABG surgery performed off-pump.
* Written informed consent to participate in this study.
* Patient and surgical procedure appropriate for treatment with either sufentanil or remifentanil.

Exclusion Criteria:

* Refusal to participate in this study.
* Age: younger than 18 years.
* Pregnant.
* BMI > 35 kg/m2.
* Patients in which atropine is contra-indicated.
* Patients in which sufentanil or remifentanil at the proposed doses are contra-indicated.
* Urgent or emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
CO | During anaesthesia

SECONDARY OUTCOMES:
MAP | During anaesthesia
Tissue oxygen saturation | During anaesthesia
CO | During anaesthesia
  CO obtained by different devices/methods (i.e. the Vigileo device and TEE)

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Poterman M, Kalmar AF, Buisman PL, Struys MMRF, Scheeren TWL. Improved haemodynamic stability and cerebral tissue oxygenation after induction of anaesthesia with sufentanil compared to remifentanil: a randomised controlled trial. BMC Anesthesiol. 2020 Oct 7;20(1):258. doi: 10.1186/s12871-020-01174-9. PMID 33028197